CLINICAL TRIAL: NCT03892577
Title: Real-world Study for Targeted Therapy and Immunotherapy in Patients With Advanced Hepatobiliary Tumors: a Multi-centers, Open-assess Observational Study.
Brief Title: Real-world Study for Patients With Advanced Hepatobiliary Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: OrigiMed (Industry)
Responsible Party: Sponsor
Other Study IDs: JS-1391
Record Dates: First submitted 2018-12-25; First posted 2019-03-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Objective Response Rate; Progression-free Survival; Overall Survival; Disease Control Rate; Duration of Response; Five-year Survival Rate; Quality of Life
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — High-Throughput Sequencing
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced hepatobiliary tumors: 2000 patients with advanced hepatobiliary tumors will be enrolled and the enroll patients should be treat with any type of the following three treatment program:
  1. Monotherapy or combination therapy with the targeted drug related to genetic variation of the subject;
  2. Treatment with pan-target anti-angiogenic drugs, such as sorafenib, regorafenib, lenvatinib, apatinib, etc;
  3. Immunotherapy or immunotherapy combined with targeted therapy or (and) chemotherapy.
  Interventions: Drug: Precision oncology including targeted therapy and immunotherapy

INTERVENTIONS:
Drug: Precision oncology including targeted therapy and immunotherapy — Therapeutic regimens are based on the clinicopathological features, genomic alterations, advices from multidisciplinary tumor board and willings from patients.

SUMMARY:
The investigators design a large sample size study in the real-world to explore whether targeted therapy and immunotherapy can improve the survival, quality of life and drug safety of patients with advanced hepatobiliary tumors, and analyze the correlation between genetic variation and the effectiveness of therapy.

DETAILED DESCRIPTION:
This trial is a multicenter, non-random, open and observational real-world study. It is estimated that 2000 patients with advanced hepatobiliary tumors will be enrolled in about 20 research centers. And it is planned to complete the enrollment within 2 years and it is expected that all enrolled subjects will reach the observation end point in 5 years.

After primary screening of all the patients, the investigators will further collect next-generation sequence(NGS) data and immunohistochemical data from the subjects, and enroll patients with any type of the following three treatment program: 1. Monotherapy or combination therapy with the targeted drug related to genetic variation of the subject; 2. Treatment with pan-target anti-angiogenic drugs, such as sorafenib, regorafenib, lenvatinib, apatinib, etc; 3. Immunotherapy or immunotherapy combined with targeted therapy.

The investigators will collect subjects' data from assessment centers each month and the efficacy, quality of life, and safety of treatment will be evaluated.

This trial plans to conduct an interim analysis and final analysis after collecting 500 cases, 1000 cases, and 2000 subjects, 3000 subjects,and explore the clinical application value of targeted therapy and immunotherapy in advanced hepatobiliary tumors in real world.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria：

1. ≥18 years old, gender is not limited, and life expectancy is at least 6 months.
2. Diagnosed as primary liver cancer or biliary malignant tumor by histopathology or confirmed by imaging as HCC (by the American Association for the Study of Liver Diseases or standard for the diagnosis and treatment of primary liver cancer 2017 in China).
3. The Barcelona staging classification: class B-C.
4. Child-Pugh classification: class A-B.
5. At least one measurable lesion (RECIST v1.1)
6. Unable to perform radical surgery or patient refuse surgery.
7. Subjects need palliative treatment, and have received or are undergoing any of the following three treatments:

   * Monotherapy or combination therapy with targeted drug associated with genetic variation in the subject.
   * Or, treat with pan-target anti-vascular drugs, such as sorafenib, regorafenib, lenvatinib, apatinib.
   * Or, immunotherapy or immunotherapy combined with targeted therapy or (and) classical chemotherapy.
8. Subjects volunteer to participate in the study and sign informed consent.

Exclusion Criteria:

Patients with one or more of the following criteria should be excluded:

1. Patients with early hepatobiliary tumor.
2. The Barcelona staging classification: class A.
3. Child-Pugh classification: class C.
4. Radical surgical resection.
5. CT or MRI shows unclear tumor boundary or no measurable lesions (RECIST v1.1).
6. Drug abuse, or any medical, psychological, or social condition that may affect the study, patient compliance, or even compromise the safety of the patient.
7. Conduct other experimental drug treatments other than this test within 4 weeks before the start of the study; or participate in another clinical study that has an impact on the results of this study.
8. Mental or medical instability makes patients unable or unwilling to sign informed consent.
9. Patients after comprehensive assessment are considered by the investigators to be unsuitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Advanced Hepatobilary Tumors.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | two years
  Time from the date of initial treatment to death for any cause.
Progression-free Survival (PFS) | six months
  A duration from the date of initial treatment with apatinib to disease progression (as defined by RECIST) or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  Percentage of subjects with complete response and partial response.
Disease Control Rate (DCR) | six months
  Percentage of subjects with complete remission, partial remission, or stable disease during treatment or within 30 days of termination of test drug.
Incidence of Treatment-Emergent Adverse Event | one year
  Percentage of subjects who develop any adverse events (CTCAE 4.0).
Quality of Life (QoL) after treatment | one year
  The life quality of every subject will be assessed every 3 months according to the 45-item FACT-Hep questionnaire, which assesses generic HRQL concerns and disease-specific issues.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, Study Chair — Chinese Academy of Medical Sciences & Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Moriguchi M, Umemura A, Itoh Y. Current status and future prospects of chemotherapy for advanced hepatocellular carcinoma. Clin J Gastroenterol. 2016 Aug;9(4):184-90. doi: 10.1007/s12328-016-0670-7. Epub 2016 Jul 11. PMID 27401471
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Sharma A, Dwary AD, Mohanti BK, Deo SV, Pal S, Sreenivas V, Raina V, Shukla NK, Thulkar S, Garg P, Chaudhary SP. Best supportive care compared with chemotherapy for unresectable gall bladder cancer: a randomized controlled study. J Clin Oncol. 2010 Oct 20;28(30):4581-6. doi: 10.1200/JCO.2010.29.3605. Epub 2010 Sep 20. PMID 20855823
- [Background] Rodriguez R, Miller KM. Unravelling the genomic targets of small molecules using high-throughput sequencing. Nat Rev Genet. 2014 Dec;15(12):783-96. doi: 10.1038/nrg3796. Epub 2014 Oct 14. PMID 25311424
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Hofstatter E, Mehra K, Yushak M, Pusztai L. Tumor profiling and the incidentalome: patient decisions and risks. Future Oncol. 2015;11(24):3299-305. doi: 10.2217/fon.15.260. Epub 2015 Nov 12. PMID 26562094
- [Background] Endrullat C, Glokler J, Franke P, Frohme M. Standardization and quality management in next-generation sequencing. Appl Transl Genom. 2016 Jul 1;10:2-9. doi: 10.1016/j.atg.2016.06.001. eCollection 2016 Sep. PMID 27668169
- [Background] Gadgeel SM. Personalized Therapy of Non-small Cell Lung Cancer (NSCLC). Adv Exp Med Biol. 2016;890:203-22. doi: 10.1007/978-3-319-24932-2_11. PMID 26703806
- [Background] Millner LM, Strotman LN. The Future of Precision Medicine in Oncology. Clin Lab Med. 2016 Sep;36(3):557-73. doi: 10.1016/j.cll.2016.05.003. PMID 27514468
- [Background] Drilon A, Wang L, Arcila ME, Balasubramanian S, Greenbowe JR, Ross JS, Stephens P, Lipson D, Miller VA, Kris MG, Ladanyi M, Rizvi NA. Broad, Hybrid Capture-Based Next-Generation Sequencing Identifies Actionable Genomic Alterations in Lung Adenocarcinomas Otherwise Negative for Such Alterations by Other Genomic Testing Approaches. Clin Cancer Res. 2015 Aug 15;21(16):3631-9. doi: 10.1158/1078-0432.CCR-14-2683. Epub 2015 Jan 7. PMID 25567908
- [Background] Li S, Mao M. Next generation sequencing reveals genetic landscape of hepatocellular carcinomas. Cancer Lett. 2013 Nov 1;340(2):247-53. doi: 10.1016/j.canlet.2012.09.027. Epub 2012 Oct 12. PMID 23063663
- [Background] Schulze K, Nault JC, Villanueva A. Genetic profiling of hepatocellular carcinoma using next-generation sequencing. J Hepatol. 2016 Nov;65(5):1031-1042. doi: 10.1016/j.jhep.2016.05.035. Epub 2016 Jun 2. PMID 27262756
- [Result] Wang YY, Yang X, Wang YC, Long JY, Sun HS, Li YR, Xun ZY, Zhang N, Xue JN, Ning C, Zhang JW, Zhu CP, Zhang LH, Yang XB, Zhao HT. Clinical outcomes of lenvatinib plus transarterial chemoembolization with or without programmed death receptor-1 inhibitors in unresectable hepatocellular carcinoma. World J Gastroenterol. 2023 Mar 14;29(10):1614-1626. doi: 10.3748/wjg.v29.i10.1614. PMID 36970591
- [Result] Yang X, Chen B, Wang Y, Wang Y, Long J, Zhang N, Xue J, Xun Z, Zhang L, Cheng J, Lei J, Sun H, Li Y, Lin J, Xie F, Wang D, Pan J, Hu K, Guan M, Huo L, Shi J, Yu L, Zhou L, Zhou J, Lu Z, Yang X, Mao Y, Sang X, Lu Y, Zhao H. Real-world efficacy and prognostic factors of lenvatinib plus PD-1 inhibitors in 378 unresectable hepatocellular carcinoma patients. Hepatol Int. 2023 Jun;17(3):709-719. doi: 10.1007/s12072-022-10480-y. Epub 2023 Feb 8. PMID 36753026
- [Result] Zhu C, Xue J, Wang Y, Wang S, Zhang N, Wang Y, Zhang L, Yang X, Long J, Yang X, Sang X, Zhao H. Efficacy and safety of lenvatinib combined with PD-1/PD-L1 inhibitors plus Gemox chemotherapy in advanced biliary tract cancer. Front Immunol. 2023 Jan 18;14:1109292. doi: 10.3389/fimmu.2023.1109292. eCollection 2023. PMID 36742297
- [Result] Xie F, Chen B, Yang X, Wang H, Zhang G, Wang Y, Wang Y, Zhang N, Xue J, Long J, Li Y, Sun H, Xun Z, Liu K, Chen X, Song Y, Yang X, Lu Z, Mao Y, Sang X, Lu Y, Zhao H. Efficacy of immune checkpoint inhibitors plus molecular targeted agents after the progression of lenvatinib for advanced hepatocellular carcinoma. Front Immunol. 2022 Dec 9;13:1052937. doi: 10.3389/fimmu.2022.1052937. eCollection 2022. PMID 36569829
- [Result] Chen B, Lei J, Zhao H, Dong J, Zeng Z, Li Y, Yu L, Zhou L, Jia A, Lu Y, Cheng J. Efficacy and Safety of TKI Plus PD-1 Inhibitors in Elderly uHCC Patients: A Retrospective Study. J Hepatocell Carcinoma. 2022 Nov 8;9:1171-1185. doi: 10.2147/JHC.S387254. eCollection 2022. PMID 36389129
- [Result] Ning C, Zhang X, Yang X, Sang X, Zhao H, Wang H. Conversion therapy of stage IVb unresectable gallbladder carcinoma. Hepatobiliary Surg Nutr. 2022 Apr;11(2):335-337. doi: 10.21037/hbsn-22-78. No abstract available. PMID 35464281
- [Result] Zuo B, Yang X, Yang X, Bian J, Long J, Wang D, Ning C, Wang Y, Xun Z, Wang Y, Lu X, Mao Y, Sang X, Zhao H. A real-world study of the efficacy and safety of anti-PD-1 antibodies plus lenvatinib in patients with advanced gallbladder cancer. Cancer Immunol Immunother. 2022 Aug;71(8):1889-1896. doi: 10.1007/s00262-021-03121-0. Epub 2022 Jan 13. PMID 35022908
- [Result] Mao J, Wang D, Long J, Yang X, Lin J, Song Y, Xie F, Xun Z, Wang Y, Wang Y, Li Y, Sun H, Xue J, Song Y, Zuo B, Zhang J, Bian J, Zhang T, Yang X, Zhang L, Sang X, Zhao H. Gut microbiome is associated with the clinical response to anti-PD-1 based immunotherapy in hepatobiliary cancers. J Immunother Cancer. 2021 Dec;9(12):e003334. doi: 10.1136/jitc-2021-003334. PMID 34873013
- [Result] Yang X, Xu H, Zuo B, Yang X, Bian J, Long J, Wang D, Zhang J, Ning C, Wang Y, Xun Z, Wang Y, Lu X, Mao Y, Sang X, Zhao H. Downstaging and resection of hepatocellular carcinoma in patients with extrahepatic metastases after stereotactic therapy. Hepatobiliary Surg Nutr. 2021 Aug;10(4):434-442. doi: 10.21037/hbsn-21-188. PMID 34430522
- [Result] Yang X, Hu Y, Yang K, Wang D, Lin J, Long J, Xie F, Mao J, Bian J, Guan M, Pan J, Huo L, Hu K, Yang X, Mao Y, Sang X, Zhang J, Wang X, Zhang H, Zhao H. Cell-free DNA copy number variations predict efficacy of immune checkpoint inhibitor-based therapy in hepatobiliary cancers. J Immunother Cancer. 2021 May;9(5):e001942. doi: 10.1136/jitc-2020-001942. PMID 33972389
- [Result] Wang DX, Yang X, Lin JZ, Bai Y, Long JY, Yang XB, Seery S, Zhao HT. Efficacy and safety of lenvatinib for patients with advanced hepatocellular carcinoma: A retrospective, real-world study conducted in China. World J Gastroenterol. 2020 Aug 14;26(30):4465-4478. doi: 10.3748/wjg.v26.i30.4465. PMID 32874058
- [Result] Lin J, Yang X, Long J, Zhao S, Mao J, Wang D, Bai Y, Bian J, Zhang L, Yang X, Wang A, Xie F, Shi W, Yang H, Pan J, Hu K, Guan M, Zhao L, Huo L, Mao Y, Sang X, Wang K, Zhao H. Pembrolizumab combined with lenvatinib as non-first-line therapy in patients with refractory biliary tract carcinoma. Hepatobiliary Surg Nutr. 2020 Aug;9(4):414-424. doi: 10.21037/hbsn-20-338. PMID 32832493
- [Derived] Yang X, Lian B, Zhang N, Long J, Li Y, Xue J, Chen X, Wang Y, Wang Y, Xun Z, Piao M, Zhu C, Wang S, Sun H, Song Z, Lu L, Dong X, Wang A, Liu W, Pan J, Hou X, Guan M, Huo L, Shi J, Zhang H, Zhou J, Lu Z, Mao Y, Sang X, Wu L, Yang X, Wang K, Zhao H. Genomic characterization and immunotherapy for microsatellite instability-high in cholangiocarcinoma. BMC Med. 2024 Jan 29;22(1):42. doi: 10.1186/s12916-024-03257-7. PMID 38281914
- [Derived] Chao J, Wang S, Wang H, Zhang N, Wang Y, Yang X, Zhu C, Ning C, Zhang X, Xue J, Zhang L, Piao M, Wang M, Yang X, Lu L, Zhao H. Real-world cohort study of PD-1 blockade plus lenvatinib for advanced intrahepatic cholangiocarcinoma: effectiveness, safety, and biomarker analysis. Cancer Immunol Immunother. 2023 Nov;72(11):3717-3726. doi: 10.1007/s00262-023-03523-2. Epub 2023 Oct 3. PMID 37787790
- [Derived] Wang Y, Zhang N, Xue J, Zhu C, Wang Y, Zhang L, Yang X, Wang H, Wang S, Chao J, Yang X, Zhao H. Safety and feasibility of toripalimab plus lenvatinib with or without radiotherapy in advanced BTC. Front Immunol. 2023 Jan 17;14:1084843. doi: 10.3389/fimmu.2023.1084843. eCollection 2023. PMID 36733485